CLINICAL TRIAL: NCT05240755
Title: Effectiveness of Cannabidiol vs. Narcotics for Post Operative Pain Control in Elective Shoulder Arthroscopic Surgery
Acronym: CBDS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Responsible Party: Principal Investigator, Michael C. Doarn, Principal Investigator, Clinical Professor of Orthopaedic Surgery - USF, Foundation for Orthopaedic Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USF003668
Record Dates: First submitted 2022-02-02; First posted 2022-02-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-09

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (No Intervention): Opioid standard of care: Tramadol 50 mg PO PRN #30, Hydrocodone/Acetaminophen 5/325 PO PRN #30
- Cannabidiol Oil 100 mg (Experimental): CBD 100 mg PO liquid suspension QD starting 30 days prior and finishing 30 days post-op
  Interventions: Drug: Cannabidiol Oil
- Cannabidiol Oil 200 mg (Experimental): CBD 200 mg PO liquid suspension QD starting 30 days prior and finishing 30 days post-op
  Interventions: Drug: Cannabidiol Oil

INTERVENTIONS:
Drug: Cannabidiol Oil — Subjects will self-administer CBD sublingually.
  Arms: Cannabidiol Oil 100 mg; Cannabidiol Oil 200 mg

SUMMARY:
This study is a prospective, randomized, nonblinded trial to evaluate the effectiveness of Cannabidiol (CBD) oil on post-operative pain control compared to opioid medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Requiring shoulder arthroscopic surgery for soft tissue pathology
* Able to complete surveys and follow-up visits

Exclusion Criteria:

* Younger than 18 years of age
* Shoulder dislocation, fracture, previous surgery, coexisting extremity pathology, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 30 days post-operatively
  Numerical Pain Scale (NRS): 0 being no pain, 10 being the worst pain imaginable. Higher scores are worse outcomes.

SECONDARY OUTCOMES:
Sleep Quality | 30 days preoperatively leading up to surgery then 30 days postoperatively as well. Outcomes will be collected from surgery to 6 weeks postoperatively.
  Insomnia Severity Index

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States